CLINICAL TRIAL: NCT06183151
Title: CApillary-VEnous Paired Collection (CAVE)
Brief Title: Capillary-Venous Paired Collection
Acronym: CaVe
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CAVE-USA
Record Dates: First submitted 2023-11-28; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Participants: All participants to undergo the same study method. Where all participants are to donate capillary blood to complete 2 tests on the investigational system and the remnant blood sample from routine CBC testing will also be tested on the investigational system. The routine CBC results will be compared to the results obtained by the investigational system.
  Interventions: Device: Entia Liberty System

INTERVENTIONS:
Device: Entia Liberty System — See arm/group description

SUMMARY:
This study is recruiting participants to donate 2 capillary blood samples to be tested on the investigational system. At the same time, remnant routine blood samples used for Complete Blood Count (CBC) testing from the same participants will be tested on the investigation system. The participants' routine CBC results analyzed on the gold standard laboratory analyzer (comparator) will be collected and compared against the results obtained from the testing of capillary blood samples and remnant blood samples on the investigational system. The participants' involvement in the study is only for the duration of collecting the blood samples. No follow-up is anticipated. The results from the investigational system is for research use only and will not inform or change the participants' treatment or care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at the time of study entry
* Currently receiving standard of care systemic anti-cancer therapy (chemotherapy, immunotherapy, endocrine and targeted therapy) for solid organ malignancy
* Scheduled to be undergoing routine CBC blood tests as part of standard of care
* Can provide written informed consent
* In the Investigator's opinion, is able and willing to comply with all study requirements

Exclusion Criteria:

* History or current diagnosis of hematological malignancy (including bone and lymph)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients undergoing treatment and attending clinic for Complete Blood Count (CBC) test
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
To validate the measurement performance of the investigational system (bias and %bias) | through study completion, estimated 6 months
  The difference between the measured parameters of the comparator and investigational system will provide the bias (and therefore also the % bias) of the investigational system, which will be checked against pre-determined acceptance criteria.
To validate the measurement performance of the investigational system (regression) | through study completion, estimated 6 months
  The plotted difference between the measured parameters of the comparator and investigational system will provide the regression, which will be checked against pre-determined acceptance criteria.
To validate the measurement performance of the investigational system (CV and SD) | through study completion, estimated 6 months
  The difference between the measured parameters of the comparator and investigational system will inform the Coefficient of Variation and Standard Deviation of the dataset, which will be checked against pre-determined acceptance criteria.